CLINICAL TRIAL: NCT04243447
Title: Identification of Predictors for Clinical Outcomes in Femoroacetabular Impingement Surgery
Acronym: DoD FAI-2
Status: Active, not recruiting | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Collaborators: San Antonio Military Medical Center (U.S. Federal Agency); Corewell Health East (Other); Boston Children's Hospital (Other); CHU de Quebec-Universite Laval (Other); Mayo Clinic (Other); Twin Cities Orthopedics (Other); Regents of the University of Michigan (Unknown); Ottawa Hospital Research Institute (Other); University of Texas Southwestern Medical Center (Other); University of Iowa (Other); University of Colorado, Denver (Other); Children's Hospital of Eastern Ontario (Other); University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: 201909174
Record Dates: First submitted 2020-01-17; First posted 2020-01-28 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Femoracetabular Impingement
Keywords: Femoracetabular Impingement (FAI); Low-dose computed tomography (CT); Patient Reported Outcomes (PROs); Academic Network for Conservational Hip Outcomes Research (ANCHOR); Hip Arthroscopy; Osteoarthritis (OA)
MeSH Terms: conditions — Femoracetabular Impingement; Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The overarching goal of the study is to improve the surgical treatment outcomes of FAI, which is affecting an increasing number of military personnel and young active individuals in the general population. The proposed study will investigate critical patient, disease, and surgical treatment predictors of FAI surgery outcomes.

DETAILED DESCRIPTION:
PROCEDURES:

Potential participants will be identified at their initial PI's outpatient clinic at which the PI will meet with the patient and determine if the patient should be treated surgically due to a diagnosis of FAI. Once the PI identifies the patient as a surgical candidate, the research study team in the clinic will approach the patient with study information to discuss. If the patient would like to participate, the patient will sign an informed consent document (assent document for minors) and begin completing study-specific information. If the patient would like to take the study documents home to consider participation, the research team member will provide his/her contact information to the patient.

SPECIFIC AIMS:

1. Determine the predictors of mid-term patient-reported outcomes (PROs) and treatment failures in an established prospective longitudinal cohort of Femoroacetabular Impingement (FAI) surgeries.
2. Determine the impact of three-dimensional femoral and acetabular morphology on PROs at short-term follow-up in a novel prospective longitudinal cohort of arthroscopic FAI surgery.
3. Determine if the new Patient-Reported Outcome Measurement Information System (PROMIS) correlates with legacy PROs in patients undergoing FAI surgery.

DATA COLLECTION:

1. Retrospective Follow-up (FAI-1): The original cohort includes previously consented participants in a closed-to-enrollment study who underwent FAI surgical treatment in the past. This cohort will be followed to investigate the most important predictors of FAI surgery outcomes. In Specific Aim 1, we propose to analyze mid-term follow-up (minimum 8 years) of the FAI-1 cohort to identify important predictors of treatment outcomes and failures in FAI surgery.
2. Prospective Enrollment (FAI-2): Consented participants, in the actively enrolling study, will be enrolled in a new multicenter longitudinal prospective arthroscopic FAI surgery cohort and followed to a minimum 2 years post-surgery (T2). The primary outcome measures will be the collection of the patient report outcomes (PROs) that will be analyzed in order to improve surgical care and outcomes. These clinical outcome metrics will be assessed at baseline, 3 months, 6 month, 1 year, and 2 year postoperatively.

ELIGIBILITY:
Inclusion Criteria:

1. Age 14 - 40 years
2. Skeletally Mature
3. Failure of 6 weeks of conservative treatment
4. Primary surgery (Hip Arthroscopic Treatment)

   a. Surgical treatment of FAI with hip arthroscopy
5. Tonnis 0 -1 OA, with greater than 2 mm of joint space
6. Clinical diagnosis of FAI (cam or combined; alpha >50 degrees)

Exclusion Criteria:

1. Not a surgical candidate
2. Skeletally Immature
3. Acetabular Dysplasia (LCEA < 20)
4. Tonnis 2+ OA
5. Previous ipsilateral hip surgery
6. Previous major hip trauma (hip fractures, hip dislocations)
7. Additional disease processes (e.g., Avascular Necrosis (AVN), synovial disease, Ehlers-Danlos Syndrome (EDS), neuromuscular disorders)
8. Unable to consent due to mental faculty
9. Pregnant women
10. Non-English speaking patients
11. Prisoners or other vulnerable populations

Ages: 14 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Skeletally mature patients being treated surgically for FAI after failing conservative treatment.
Sampling Method: Non-Probability Sample
Enrollment: 747 (Actual)
Dates: Start 2020-02-02 (Actual); Primary Completion 2025-11-29 (Estimated); Study Completion 2025-11-29 (Estimated)

PRIMARY OUTCOMES:
Hip disability and Osteoarthritis Outcome Score (HOOS) | Pre operative (Baseline), change from baseline HOOS at 3 months, change from baseline HOOS at 6 months, change from baseline HOOS at 1 year, and change from baseline HOOS at 2 year.
  HOOS is a questionnaire constructed to assess patient-relevant outcomes in five separate sub-scales (pain, symptoms, activity of daily living, sport and recreation function and hip-related quality of life). HOOS is scored 0-100 with higher scores being the best outcome.
Short Form Health Survey (SF-12) | Pre operative (Baseline), change from baseline SF-12 at 3 months, change from baseline SF-12 at 6 months, change from baseline SF-12 at 1 year, and change from baseline SF-12 at 2 year
  The SF-12 is a shortened, validated, patient-reported survey of patient health with questions pulled directly from the longer form SF-36. SF-12 is scored 0-100 with higher scores being the best outcome.
Patient-Reported Outcomes Measurement Information System (PROMIS) - Pain Interference (PI) | Pre operative (Baseline), change from baseline PROMIS - PI at 3 months, change from baseline PROMIS - PI at 6 months, change from baseline PROMIS -PI at 1 year, and change from baseline PROMIS - PI at 2 year
  PROMIS is a set of person-centered measures that evaluates and monitors physical, mental, and social health in adults and children. It can be used with the general population and with individuals living with chronic conditions. This specific PROMIS survey assesses a patient's pain interference. PROMIS - PI is scored from 38.7-83.8 with the lower scores being the best outcome.
Patient-Reported Outcomes Measurement Information System (PROMIS) - Physical Function (PF) | Pre operative (Baseline), change from baseline PROMIS - PF at 3 months, change from baseline PROMIS - PF at 6 months, change from baseline PROMIS -PF at 1 year, and change from baseline PROMIS - PF at 2 year
  PROMIS is a set of person-centered measures that evaluates and monitors physical, mental, and social health in adults and children. It can be used with the general population and with individuals living with chronic conditions. This specific PROMIS survey assesses a patient's physical function. PROMIS - PF is scored from 14.7-75.6 with the higher scores being the best outcome.
Patient-Reported Outcomes Measurement Information System (PROMIS) - Mobility (M) | Pre operative (Baseline), change from baseline PROMIS - M at 3 months, change from baseline PROMIS - M at 6 months, change from baseline PROMIS -M at 1 year, and change from baseline PROMIS - M at 2 year
  PROMIS is a set of person-centered measures that evaluates and monitors physical, mental, and social health in adults and children. It can be used with the general population and with individuals living with chronic conditions. This specific PROMIS survey assesses a patient's mobility. PROMIS - M is scored from 18.2-60.2 with the higher scores being the best outcome.
Patient-Reported Outcomes Measurement Information System (PROMIS) - Depression (D) | Pre operative (Baseline), change from baseline PROMIS - D at 3 months, change from baseline PROMIS - D at 6 months, change from baseline PROMIS - D at 1 year, and change from baseline PROMIS - D at 2 year
  PROMIS is a set of person-centered measures that evaluates and monitors physical, mental, and social health in adults and children. It can be used with the general population and with individuals living with chronic conditions. This specific PROMIS survey assesses a patient's depression. PROMIS - D is scored from 34.2-84.4 with the lower scores being the best outcome.
Patient-Reported Outcomes Measurement Information System (PROMIS) - Anxiety (A) | Pre operative (Baseline), change from baseline PROMIS - A at 3 months, change from baseline PROMIS - A at 6 months, change from baseline PROMIS - A at 1 year, and change from baseline PROMIS - A at 2 year
  PROMIS is a set of person-centered measures that evaluates and monitors physical, mental, and social health in adults and children. It can be used with the general population and with individuals living with chronic conditions. This specific PROMIS survey assesses a patient's anxiety. PROMIS - A is scored from 32.9-84.9 with the lower scores being the best outcome.

SECONDARY OUTCOMES:
University of California Los Angeles Activity Score (UCLA Score) | Pre operative (Baseline), change from baseline UCLA Score at 3 months, change from baseline UCLA Score at 6 months, change from baseline UCLA Score at 1 year, and change from baseline UCLA Score at 2 year
  UCLA Score represents a reliable tool for assessing the level of physical activity and the return to sport high functional demand after hip surgery. The UCLA Score is scored from 0-10 with higher scores being the best outcome.
International Hip Outcome Tool (iHot-12) | Pre operative (Baseline), change from baseline iHOT-12 at 3 months, change from baseline iHOT-12 at 6 months, change from baseline iHOT-12 at 1 year, and change from baseline iHOT-12 at 2 year
  iHOT-12 is a validated 12-item short form of iHot-33. It was designed to measure the impact of hip disease in young, active patients and to measure the effect of treatment of this disease.
Modified Harris Hip Score (mHHS) | Pre operative (Baseline), change from baseline mHHS at 3 months, change from baseline mHHS at 6 months, change from baseline mHHS at 1 year, and change from baseline mHHS at 2 year
  The mHHS is a reliable and valid tool for assessment of functional outcome, post total hip replacement in Indian patients, with a positive correlation with the standard Harris Hip Score. mHHS is scored 0-100 with higher scores being the best outcome.
Brief Resilience Scale (BRS) | Pre operative (Baseline)
  The BRS was created to assess the ability to bounce back or recover from stress.
Mobility, Stability, and Pain (MSP Question) | Pre operative (Baseline), 3 months, 6 month
  Outcome measure to assess a patient's greatest issue with their hip. Asks a patient to rank mobility, stability, and pain from biggest problem to least problem.

CONTACTS AND LOCATIONS:
Overall Officials: John C Clohisy, MD, Principal Investigator — Washington University School of Medicine
Locations (13):
- United States (10):
  - University of Colorado, Aurora, Colorado
  - University of Iowa, Iowa City, Iowa
  - Boston Children's Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Twin Cities Orthopedics, Edina, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Scottish Rite Hospital for Children, Dallas, Texas
  - San Antonio Military Medical Center, San Antonio, Texas
  - University of Wisconsin, Madison, Madison, Wisconsin
- Canada (3):
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - CHU de Quebec - Universite Laval, Québec, Quebec

DOCUMENTS (1):
  • Informed Consent Form (2020-06-09): https://cdn.clinicaltrials.gov/large-docs/47/NCT04243447/ICF_000.pdf